CLINICAL TRIAL: NCT02899117
Title: Pilot Yoga Intervention to Improve Pediatric Cancer Patients' Sleep & Life Quality and Parents' Well-Being
Brief Title: Yoga Intervention to Improve Pediatric Cancer Patients' Sleep & Life Quality and Parents' Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Andrea Orsey, Assitant Professor Dept of Hematology Oncology, Connecticut Children's Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pilot Yoga 1
Record Dates: First submitted 2016-08-23; First posted 2016-09-14 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yoga intervention (Experimental): Patients in the yoga intervention group will have 4 yoga sessions with a certified yoga instructor while they are in the cancer clinic or on the inpatient floor.
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — There are 4 yoga sessions completed with a certified instructor during cancer treatment

SUMMARY:
The proposed project will examine feasibility and preliminary efficacy of a yoga intervention in the pediatric oncology unit at Connecticut Children's Medical Center (CCMC) and includes two parts: (1) a survey of children and parents regarding preferences (e.g., convenient days/times), experiences and expectations regarding yoga (including barriers and positive expectancies) and (2) an eight week clinical trial of a yoga intervention in 10 pairs of children and parents.

DETAILED DESCRIPTION:
The specific aims and hypotheses for this seed grant are to collect and assess data on:

Aim 1 feasibility - perceived barriers/solutions, interest and accrual rates, attendance per session, participant retention, evidence of institutional support and resource commitment Hypothesis 1: A yoga intervention is feasible among pediatric oncology patients and their parents; (2) preliminary efficacy - including effect sizes for calculating power Hypothesis 2a: A yoga intervention improves pediatric oncology patients' fatigue, QOL, and sleep.

Hypothesis 2b: A yoga intervention improves parental QOL and caregiver burden.

We will be using the following questionnaires and scales to help answer the quesitons related to the hypotheses and aims:

PedsQL 4.0 PedsQL 3.0 Cancer Module The Fatigue Scale SleepDiary Actigraphy data. Child Home Yoga Practice Diary Satisfaction survey

Questionnaires noted below are given only to the parents:

SF-12 Zarit Caregiver Burden Index Yoga Satisfaction Survey

Study participants will have 4 yoga sessions and the questionnaires and surveys are done prior to the first yoga session and after the last yoga session.

The yoga sessions are created with both the study participant and a certified yoga instructor. The patients are given the yoga routine to practice at home at their leisure.

ELIGIBILITY:
Inclusion Criteria:

* Parents and children (ages 8-18) undergoing treatment (chemotherapy and/or radiation therapy) for cancer.
* Cancer diagnosis, between the ages of 8-18 year, English speaking, and medically cleared to participate in yoga.
* Parents will be eligible if they are over 18 years old, English speaking, and physically able to participate in yoga.

Exclusion Criteria:

* Children and parents not meeting inclusion criteria

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2014-08; Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of yoga intervention, perceived barriers/solutions | Change from baseline barriers/solutions at 8 weeks post baseline visit
  The data will be assessed on perceived barriers/solutions.
Assess level of interest utlizing data from the Yoga satisfaction survey | Data collected at baseline and 8 weeks post baseline visit
  Data will be assessed by level of interest utilizing data from the yoga satisfcation survey. Most responses will be on a Likert scale while some specific questions will be other formats (i.e. open ended questions). These questions will help to inform the intervention.
Feasibility of yoga intervention, assessed by study accrual rates | Baseline and 8 weeks post baseline visit
  Data will be assessed by accrual rates
Feasibility of yoga intervention, assessed by study visit attendance | Baseline and 8 weeks post baseline visit
  Data will be assessed by study visit attendance
Feasibility of yoga intervention, assessed by study patient retention | Baseline and 8 weeks post baseline visit
  Data will be assessed by the number of patients who remain in the study
Feasibility of yoga intervention, assessed by institutional support | Baseline and 8 weeks post baseline visit
  Data will be reviewed for evidence of institutional support
Feasibility of yoga intervention, assessed by institutional commitment of resources. | Assessments are collected at baseline and 8 weeks post baseline visit
  Data will be reviewed for institutional resource commitment

SECONDARY OUTCOMES:
Improvement in sleep of Patient | Assessments are collected at baseline and 8 weeks post baseline visit
  Sleep will be assessed via diary of sleep and actigraphy
Improvement in quality of life Patient | Assessments are collected at baseline and 8 weeks post baseline visit
  Quality of life will be assessed by PedsQL 4.0 and PedsQL 3.0 Cancer Module.
Improvement in fatigue of Patient | Assessments are collected at baseline and 8 weeks post baseline visit
  Fatigue will be assessed by the Fatigue Scale (FS). The Fatigue Scale for children (FS-C) between 8-12 years and the Fatigue Scale for adolescent (FS-A) between 13-18 years.
Improvement in quality of life of Parent | Assessments are collected at baseline and 8 weeks post baseline visit
  Parent quality of life will be assessed by the SF-12.
Improvement in caregiver burden of Parent. | Assessments are collected at baseline and 8 weeks post baseline visit
  Caregiver burden will be assessed by the Zarit Caregiver Burden Index

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Orsey, MD, Principal Investigator — Connecticut Childrens Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No